CLINICAL TRIAL: NCT01668602
Title: Cortical and Spinal Correlates of Post-stroke Gait Rehabilitation
Brief Title: Stroke Gait Rehabilitation Using Functional Electrical Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); American Heart Association (Other)
Responsible Party: Principal Investigator, Trisha Kesar, PT, PhD, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00058363; 5K01HD079584-02 (NIH); 13SDG13320000 (Other: American Heart Association)
Record Dates: First submitted 2012-08-15; First posted 2012-08-20 (Estimated); Results first posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Cerebrovascular Accident
Keywords: Rehabilitation; Gait disorders; Chronic stroke
MeSH Terms: conditions — Stroke; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: Assignment to either Cohort 1 or Cohort 2 will occur simultaneously and will be based on the lab/personnel and subject schedules. Participants in Cohort 1 receive only FastFES. Participants in Cohort 2 will receive 3 sessions of FastFES and 3 sessions of fast walking without FES.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Cohort 1 - FastFES Training (Experimental): Participants with chronic stroke in Cohort 1 will receive 18 training sessions of FastFES (fast treadmill walking with electrical stimulation).
  Interventions: Device: Fast Walking with Fast Functional Electrical Stimulation (FES) Training
- Cohort 2 - FastFES and Fast Walking (Experimental): Participants with chronic stroke in Cohort 2 who complete 3 sessions of FastFES and 3 sessions of fast walking.
  Interventions: Device: Fast Walking with Fast Functional Electrical Stimulation (FES) Training; Other: Fast Walking

INTERVENTIONS:
Device: Fast Walking with Fast Functional Electrical Stimulation (FES) Training — Functional electrical stimulation (FES) is a technique that causes a muscle to contract through the use of an electrical current. The therapist applies an electrical current to either the skin over the nerve, or over the bulk of the muscle, and this will cause a muscle contraction. The FES is delivered to 2 muscle groups (dorsiflexor and plantarflexor) timed appropriately with the gait cycle. FastFES gait training sessions may comprise up to six 6-minute bouts of walking with rest breaks between bouts (total 30-minutes of walking). The last training bout (bout 6) may comprise 6-minutes of over ground walking, during which subjects will be asked to walk as fast as they can. For safety, a physical therapist will walk with and guard the subject during over ground walking.
  Other Names: FastFES
Other: Fast Walking — Fast walking training sessions will be similar to FastFES in duration, dosage, structure but no FES will be provided.
  Arms: Cohort 2 - FastFES and Fast Walking

SUMMARY:
The study is a prospective interventional study to assess the changes in corticospinal excitability and spinal reflex excitability of in response to rehabilitative strategies and protocols that are commonly used during physical therapy treatment of gait disorders among post-stroke subjects. As part of this protocol, 55 individuals with chronic stroke will be assigned to either Cohort 1 or Cohort 2, and will participate in 1-18 gait training sessions. If interested, study participants can also complete both study cohorts sequentially (with at least 3-weeks duration between switching from one cohort to the second). The study examines the effects among two cohorts of post stroke patients. Cohort 1 will participate in 18 sessions of fast treadmill walking plus Functional Electrical Stimulation (FastFES) and Cohort 2 will participate in 1-3 sessions of FastFES and fast walking without FES.

DETAILED DESCRIPTION:
Stroke is the number one cause of disability. Difficulty with walking affects most stroke survivors. Walking deficits (e.g. reduced ankle flexion during swing phase, decreased forward propulsion during terminal stance) can cause risks of falls, slow walking speed, increased effort of walking, and difficulties with activities of daily living. Restoration of walking ability can improve quality of life, and is perceived as a major goal of rehabilitation by stroke survivors. Examples of interventions that are used to rehabilitate walking post-stroke are functional electrical stimulation, fast treadmill walking, and bio- feedback. While recent research has focused on comparing the effectiveness of different gait rehabilitation interventions, the neural and biomechanical mechanisms underlying different gait rehabilitation strategies are unknown. FastFES is a novel gait training intervention that combines the beneficial effects of two independent interventions: Fast treadmill walking and FES. The FastFES intervention incorporates principles of physiology, biomechanics, motor control and learning, and predictions of forward-dynamic gait simulations to improve post-stroke gait.

The overall purpose of this protocol is to assess the biomechanical and neurophysiologic effects of rehabilitative strategies and protocols that are commonly used during physical therapy treatment of gait disorders post-stroke among two cohorts of people. Aim 1 of the study will assess the changes in gait biomechanics, corticospinal excitability, and walking function during 18 sessions of gait retraining, with participants in Cohort 1. Aim 2 of the study assesses the effect of parameters such as walking speed (slow, fast, variable, split-belt walking), functional electrical stimulation parameters (short-term changes induced by fast versus FastFES, stimulation intensity, number of muscles stimulated), and bio-feedback on within-session changes in gait biomechanics, walking function, and corticospinal excitability, among participants in Cohort 2.

Within Cohort 1, participants will receive identical treatment throughout the 18 training sessions (i.e. FastFES training). Within Cohort 2, participants will participate in 3 training sessions of both FastFES and fast walking training, with a 3-week break between the two types of training.

ELIGIBILITY:
Inclusion Criteria:

* Chronic stroke (>6 months post stroke)
* First (single) lesion
* Able to walk with or without the use of a cane or walker
* Sufficient cardiovascular health and ankle stability to walk for 6 minutes at a self-selected speed without an orthoses
* Resting heart rate 40-100 beats per minute
* Resting blood pressure between 90/60-70/90

Exclusion Criteria:

* Evidence of moderate/ severe chronic white matter disease or cerebellar stroke on MRI
* Cerebellar signs (ataxic ("drunken") gait or decreased coordination during rapid alternating hand or foot movements
* Insulin dependent diabetes
* History of lower extremity joint replacement
* Score of >1 on question 1b and >0 on question 1c on NIH Stroke Scale
* Inability to communicate with investigators
* Neglect/hemianopia, or unexplained dizziness in last 6 months
* Neurologic conditions other than stroke
* Orthopedic problems in the lower limbs or spine (or other medical conditions) that limit walking
* Contraindications to transcranial magnetic stimulation (TMS) are: history of seizures, metal implants in the head or face, history of recurring or severe headaches/migraine, headache within the past 24 hours, presence of skull abnormalities or fractures, hemorrhagic stroke, history of dizziness, syncope, nausea, or loss of consciousness in the past 12 months

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trisha Kesar, PT, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allen JL, Ting LH, Kesar TM. Gait Rehabilitation Using Functional Electrical Stimulation Induces Changes in Ankle Muscle Coordination in Stroke Survivors: A Preliminary Study. Front Neurol. 2018 Dec 20;9:1127. doi: 10.3389/fneur.2018.01127. eCollection 2018. PMID 30619077

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began in August 2013 and all study follow up was completed on May 1, 2019.
Groups:
- Cohort 1 - FastFES Training: Participants with chronic stroke in Cohort 1 will receive 18 training sessions of fast walking on a treadmill plus Functional Electrical Stimulation (FastFES).
- Cohort 2 - FastFES and Fast Walking: Participants with chronic stroke in Cohort 2 who complete 3 sessions of FastFES and 3 sessions of fast walking on a treadmill.
Period: Overall Study
Arm/Group | Cohort 1 - FastFES Training | Cohort 2 - FastFES and Fast Walking
Started | 2 | 22
Cohort 2 - Began FastFES Sessions | 0 (This milestone does not apply to Cohort 1.) | 20
Cohort 2 - Completed 3 Sessions of FastFES | 0 (This milestone does not apply to Cohort 1.) | 19
Cohort 2 - Began Fast Walking Sessions | 0 (This milestone does not apply to Cohort 1.) | 20
Cohort 2 - Completed 3 Sessions of Fast Walking | 0 (This milestone does not apply to Cohort 1.) | 18
Completed | 2 | 18
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1 - FastFES Training: Participants in Cohort 1 will receive 18 training sessions of FastFES (fast treadmill walking with electrical stimulation).
- Cohort 2 - FastFES and Fast Walking: Participants in Cohort 2 who complete 3 sessions of FastFES and 3 sessions of fast walking.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - FastFES Training | Cohort 2 - FastFES and Fast Walking | Total
Number analyzed (Participants) | 2 | 22 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 12 | 13
  >=65 years | 1 | 10 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 10 | 12
  Male | 0 | 12 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 22 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Motor Evoked Potentials (MEP) Amplitude Measure in milliVolt (mV) of FastFES Versus Fast Walking After 3 Training Sessions in Cohort 2
Description: Change from baseline in MEP amplitude (transverse abdominal (TA) muscle) is used as a measure of corticospinal excitability that is assessed using a non-invasive technique called transcranial magnetic stimulation (TMS). Electrical activity from muscles in response to the TMS will be collected using surface electromyography (EMG) sensors attached to muscles that play critical roles during FastFES versus Fast walking. TMS will be delivered using two Magstim 200 stimulators connected via a BiStim module. An average of 10 TMS-evoked MEP responses will be used to comparing mean peak-to-peak MEP amplitudes in response to suprathreshold TMS delivered to the hotspot.
Time Frame: Baseline, week 3 (after 3 sessions of one intervention), week 6 (after 3 sessions of the other intervention)
Population: This analysis includes participants in Cohort 2 who had complete data for this assessment. There were issues with data collection during the training sessions and stimulus artifact causing noise in data, resulting in incomplete data for some participants.
Measure: Mean (Standard Deviation); unit: mV
Groups:
- Three Sessions of FastFES: Cohort 2 participants after having three sessions of FastFES
- Three Sessions of Fast Walking: Cohort 2 participants after having three sessions of Fast Walking
Arm/Group | Three Sessions of FastFES | Three Sessions of Fast Walking
Number analyzed (Participants) | 12 | 12
mV | 0.058 (0.110) | 0.013 (0.200)

2. Primary Outcome: Change in H-Reflex /M-Wave (Hmax/Mmax) Ratio Among FastFES Versus Fast Walking After 3 Training Sessions in Cohort 2
Description: Change from baseline in (Hmax/Mmax) ratio is used as a measure of spinal reflex excitability, that is assessed using peripheral electrical stimulation delivered to the nerves innervating the ankle muscles. An electrical stimulation electrode is placed just above the knee, and used as the anode for tibial nerve stimulation. Electrical stimulation is delivered via surface electrodes in a static position to the popliteal fossa. The subject's EMG activity will be recorded while the cathode is moved at the back of the knee to determine the location that provides the best EMG response (H-reflex). EMG activity will be recorded while 50-60 electrical stimuli (short 1 ms square pulses, ranging in intensity in milliAmpere(mA) 1-80), 7-10 seconds apart, are delivered to the muscle. Also 5-20 electrical stimulus pulses at intensities are delivered that elicit a percentage of the maximum reflex response.
Time Frame: Baseline, week 3 (after 3 sessions of one intervention), week 6 (after 3 sessions of the other intervention)
Population: This analysis includes participants in Cohort 2 who have complete data for this assessment. There were issues with data collection during the training sessions and stimulus artifact causing noise in data, resulting in incomplete data for some participants.
Measure: Mean (Standard Deviation); unit: percentage of Hmax/Mmax
Arm/Group | Three Sessions of FastFES | Three Sessions of Fast Walking
Number analyzed (Participants) | 12 | 12
percentage of Hmax/Mmax | 4.14 (0.05) | 0.44 (0.09)

3. Primary Outcome: Change in Motor Evoked Potentials (MEP) Amplitude Measure in milliVolt (mV) of FastFES After 18 Training Sessions in Cohort 1
Description: Change from baseline in MEP amplitude (TA muscle in a resting state) is used as a measure of corticospinal excitability that is assessed using a non-invasive technique called transcranial magnetic stimulation (TMS). Electrical activity from muscles in response to the TMS will be collected using surface electromyography (EMG) sensors attached to muscles that play critical roles during FastFES versus Fast walking. TMS will be delivered using two Magstim 200 stimulators connected via a BiStim module. An average of 10 TMS-evoked MEP responses will be used to comparing mean peak-to-peak MEP amplitudes in response to suprathreshold TMS delivered to the hotspot.
Time Frame: Baseline and up to 6 weeks
Population: This analysis includes participants in Cohort 1.
Measure: Mean (Standard Deviation); unit: mV
Groups:
- FastFES Training: Participants in Cohort 1 receiving 18 sessions of FastFES Training.
Arm/Group | FastFES Training
Number analyzed (Participants) | 2
mV | -0.02 (0.07)

4. Primary Outcome: Change in H-Reflex /M-Wave (Hmax/Mmax) Ratio Among FastFES Versus Fast Walking After 18 Training Sessions in Cohort 1
Description: as for outcome 2
Time Frame: Baseline and up to 6 weeks
Population: This analysis includes participants from Cohort 1.
Measure: Mean (Standard Deviation); unit: percentage of Hmax/Mmax
Arm/Group | FastFES Training
Number analyzed (Participants) | 2
percentage of Hmax/Mmax | 24.49 (45.88)

5. Secondary Outcome: Change in Peak Anterior Ground Reaction Force (AGRF) of FastFES Versus Fast Walking After 3 Training Sessions in Cohort 2
Description: Change from baseline in peak AGRF during treadmill walking will be collected using a treadmill instrumented with two force platforms under each belt. Motion analysis data will be collected during 15- to 40-second long dynamic walking trials as subjects walk on a treadmill.
Time Frame: Baseline, week 3 (after 3 sessions of one intervention), week 6 (after 3 sessions of the other intervention)
Population: This analysis includes participants from Cohort 2 who had complete data for this assessment. There were issues with data collection during the training sessions and stimulus artifact causing noise in data, resulting in incomplete data for some participants.
Measure: Mean (Standard Deviation); unit: Newtons.milliseconds (N.ms)
Arm/Group | Three Sessions of FastFES | Three Sessions of Fast Walking
Number analyzed (Participants) | 12 | 12
Newtons.milliseconds (N.ms) | 8.68 (11.76) | -2.00 (12.76)

6. Secondary Outcome: Change in Peak Anterior Ground Reaction Force (AGRF) of FastFES Versus Fast Walking After 18 Training Sessions in Cohort 1
Description: as for outcome 5
Time Frame: Baseline and up to 6 weeks
Population: This analysis includes participants in Cohort 1.
Measure: Mean (Standard Deviation); unit: Newtons.milliseconds (N.ms)
Arm/Group | FastFES Training
Number analyzed (Participants) | 2
Newtons.milliseconds (N.ms) | 15.40 (10.82)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the training sessions, from the start of the study intervention session through the last session (up to 6 weeks).
Description: In Cohort 2 there were 20 participants who received at least one session of FastFES and 19 who received at least one session of Fast Walking.
Groups:
- Cohort 1 - 18 Sessions of FastFES Training: Participants in Cohort 1 will receive 18 training sessions of FastFES (fast treadmill walking with electrical stimulation).
- Cohort 2 - Three Sessions of FastFES: Participants in Cohort 2 during training sessions of FastFES.
- Cohort 2 - Three Sessions of Fast Walking: Participants in Cohort 2 during training sessions of Fast Walking.
Arm/Group | Cohort 1 - 18 Sessions of FastFES Training | Cohort 2 - Three Sessions of FastFES | Cohort 2 - Three Sessions of Fast Walking
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/2 | 0/20 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - 18 Sessions of FastFES Training (N=2) | Cohort 2 - Three Sessions of FastFES (N=20) | Cohort 2 - Three Sessions of Fast Walking (N=20)
Lightheadedness during H-reflex evaluation (General disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/02/NCT01668602/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT01668602/Prot_SAP_001.pdf